CLINICAL TRIAL: NCT04016766
Title: Mobile Application Intervention Targeting the High Risk Drinking Practice of Prepartying
Brief Title: Brief Mobile Intervention for Prepartying
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RAND (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34AA025968 (NIH)
Record Dates: First submitted 2019-07-10; First posted 2019-07-11 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Heavy Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prepartying mobile app intervention (Experimental): Mobile app intervention
  Interventions: Behavioral: Mobile app prepartying intervention
- Control (No Intervention): Control participants receive a personalized attention control task (i.e., listing and ranking favorite movies, music, and books), which controls for the time needed by the intervention group to view the intervention material.

INTERVENTIONS:
Behavioral: Mobile app prepartying intervention — The intervention is comprised of a theoretically-informed and empirically-supported, brief, accessible, and personalized intervention to address prepartying drinking. the prepartying intervention app will be tailored toward an individual's personal goals, beliefs (perceptions, expectancies, self-efficacy), and behavior (protective strategies), and focus on the core components of brief interventions that have been cited as constructs that mediate the effects of multiple component intervention programs (e.g., correcting perceived norms, use of protective behavioral strategies, increased self-efficacy, challenging expectancies, feedback on blood alcohol level).
  Arms: Prepartying mobile app intervention

SUMMARY:
The primary objective of the research study is to develop and test a prepartying (aka "pregaming") specific brief mobile app intervention that is intended to help college students reduce their prepartying drinking behavior. Such behavior has been identified as a major contributor to alcohol-related negative consequences among young people. The investigators will first develop the intervention content based on theory and research supporting mechanisms of change in brief interventions with college students and document normative drinking information from 500 college students for inclusion in the intervention content. Investigators will then beta test the intervention with a sample of 14 heavy drinking college students. Focus group feasibility and acceptability feedback will inform the final intervention content. Investigators will then pilot test the mobile-based intervention in a randomized controlled trial of 500 college students who preparty frequently (n = 250 intervention, n = 250 attention control) and determine the efficacy of the intervention on (1) preventing heavy consumption levels during and after prepartying and on (2) reducing students' global levels of heavy drinking and consequences one and three months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* full time undergraduate college student
* between the ages of 18 and 24
* report typically prepartying at least once per week

Exclusion Criteria:

* not meeting inclusion criteria

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Prepartying frequency | Past month (30 days)
  Number of days reported prepartying on the timeline followback
Drinks during prepartying | Past month (30 days)
  Average number of drinks reported during prepartying on the timeline followback
Drinking frequency | Past month (30 days)
  Number of days reported any drinking on the timeline followback
Drinks on drinking days | Past month (30 days)
  Average number of drinks reported during drinking days on the timeline followback
21-item Brief Young Adult Alcohol Consequences Questionnaire | Past month (30 days)
  Number of 21 assessed alcohol consequences experienced (yes/no). Yes responses are summed to yield a score on this measure. Higher scores indicate experience of a greater number of consequences. Scores range from 0 (no consequences) to 21 (experience of all 21 consequences)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pedersen ER, Hummer JF, Davis JP, Fitzke RE, Tran DD, Witkiewitz K, Clapp JD. A mobile-based pregaming drinking prevention intervention for college students: A pilot randomized controlled trial. Psychol Addict Behav. 2023 Nov;37(7):841-852. doi: 10.1037/adb0000925. Epub 2023 Apr 13. PMID 37053413
- [Derived] Pedersen ER, Hummer JF, Davis JP, Fitzke RE, Christie NC, Witkiewitz K, Clapp JD. A mobile-based pregaming drinking prevention intervention for college students: study protocol for a randomized controlled trial. Addict Sci Clin Pract. 2022 Jun 18;17(1):31. doi: 10.1186/s13722-022-00314-5. PMID 35717303